CLINICAL TRIAL: NCT06297720
Title: Safety and Feasibility of Early Oral Hydration After Video-assisted Thoracoscopic Surgery: A Prospective, Randomized, and Controlled Study
Brief Title: Early Oral Hydration After Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2401110013
Record Dates: First submitted 2024-02-05; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia; Intubation Complication
Keywords: Early oral hydration; Sore throat
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hydration (Experimental): wet swab-ice cube-small amount of water
  Interventions: Behavioral: Oral hydration
- No hydration (No Intervention): According to routine care, no oral fluid supplementation is provided.

INTERVENTIONS:
Behavioral: Oral hydration — * Researchers moisten the patient's throat with a wet cotton swab. If no nausea or vomiting occurs after five minutes, proceed to the next stage.
  * Provide an ice cube of potable water for the patient to hold in their mouth. If no nausea or vomiting occurs after ten minutes, proceed to the next stage.
  * Offer 10-20ml of potable water for the patient to drink under medical supervision. If no nausea or vomiting occurs and the patient requests more water, administer 10-20ml every ten minutes, assessing for any adverse effects each time. The total water intake should not exceed 500ml.
  Arms: Oral hydration

SUMMARY:
The goal of this clinical trial is to learn about the safety and feasibility of early oral hydration in patients receiving video-assisted thoracoscopic surgery after general anesthesia. The main questions aims to answer:

* the safety and feasibility of oral hydration supplementation in the recovery room following general anesthesia.
* the degree of improvement in sore throat and dry mouth after oral hydration.
* the side effects and risks of oral hydration supplementation, such as the incidence of postoperative nausea and vomiting.
* the impact of oral hydration supplementation in the recovery room following general anesthesia on hemodynamics.
* patient satisfaction with oral hydration supplementation in the recovery room following general anesthesia.

Participants will receive a series of oral hydration from swab moistening, and ice cube hydration to water hydration in the recovery room. Researchers will compare with the standard, no-hydration group to see if it is safe and feasible to hydrate patients in the recovery room.

DETAILED DESCRIPTION:
Anesthesiologists assess the removal of the endotracheal tube post-surgery and the patient is then transferred to the recovery room for rest. The principal investigator will evaluate the consciousness status and risk of nausea and vomiting to confirm eligibility for the trial. Subsequently, the following grouping will be conducted:

1. Experimental group

   * First, moisten the patient's throat with a cotton swab dipped in water. If no nausea or vomiting occurs after five minutes, proceed to the next stage.
   * Provide an ice cube for the patient to hold in their mouth. If no nausea or vomiting occurs after ten minutes, proceed to the next stage.
   * Offer 10-20ml water for the patient to drink under medical supervision. If no nausea or vomiting occurs and the patient requests more water, administer 10-20ml of water every ten minutes, assessing for any adverse effects each time. The total water intake should not exceed 500ml.
2. Comparison group - standard care without any intervention

Evaluate the level of throat pain using VAS (Visual Analogue Scale) score, the incidence, timing, frequency of post-operative nausea and vomiting, the level of mouth dryness, the satisfaction of patients in recovery room, and the vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 70.
* Anesthesia physical status classification III or below
* Body Mass Index 30 or below
* Elective video-assisted thoracoscopic surgery

Exclusion Criteria:

* Pre-operative throat pain
* Impaired mental status
* Tendency to choke (inc. dysphagia, stroke hx.)
* Nil Per Os (NPO) less than 8 hours
* Pregnancy
* Nausea and vomiting in Operating room or Post-anesthesia care unit

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
sore throat level by VAS (Visual Analogue Scale) | From patient arrived at the PACU (Postanesthesia Care Unit) to patient being discharged, about 1-3 hours
  sore throat level by VAS (Visual Analogue Scale) measured by 0-10 point-scale
Mouth dryness | From patient arrived at the PACU (Postanesthesia Care Unit) to patient being discharged, about 1-3 hours
  Modified Schirmer tear strip test

SECONDARY OUTCOMES:
post-operative nausea and vomiting (PONV) | From patient been sent to PACU (Postanesthesia Care Unit) until discharge, about 1-3 hours
  PONV exist or not
timing of post-operative nausea and vomiting (PONV) | From patient been sent to PACU (Postanesthesia Care Unit) until discharge, about 1-3 hours
  PONV or not, if yes, record timing
duration of post-operative nausea and vomiting (PONV) | From patient been sent to PACU (Postanesthesia Care Unit) until discharge, about 1-3 hours
  PONV or not, if yes, record duration
management of post-operative nausea and vomiting (PONV) | From patient been sent to PACU (Postanesthesia Care Unit) until discharge, about 1-3 hours
  PONV or not, if yes, record management
Heart Rate in PACU (Postanesthesia Care Unit) | From patient been sent to PACU (Postanesthesia Care Unit) until discharge in every 5 minutes, about 1-3 hours
  Heart Rate (/min) in PACU (Postanesthesia Care Unit)
Blood pressure in PACU (Postanesthesia Care Unit) | From patient been sent to PACU (Postanesthesia Care Unit) until discharge in every 5 minutes, about 1-3 hours
  Blood pressure (mmHg) in PACU (Postanesthesia Care Unit)
Patient's satisfaction | Through study completion, before patients leaving PACU (Postanesthesia Care Unit)
  Patient's satisfaction measured by Likert scale (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: JUN-YU CHEN, Study Chair — +886937020809
Locations (1):
- ChangGung MH, Taoyuan District, Taiwan